CLINICAL TRIAL: NCT05365516
Title: Medical Safety Huddles - a Multi-site QI (Quality Improvement) Project
Brief Title: Medical Safety Huddles - a Multi-site QI Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sinai Health System (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 19-6357
Record Dates: First submitted 2022-04-20; First posted 2022-05-09 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Patient Safety
Keywords: Quality Improvement; Patient Safety; Physician Engagement; Huddles

STUDY DESIGN:
Intervention Model Description: The multi-centre QI project will use a stepped wedge cluster randomized design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Safety Huddles - Pre-implementation (No Intervention)
- Medical Safety Huddles - Post-implementation (Experimental)
  Interventions: Other: Implementing medical safety huddles

INTERVENTIONS:
Other: Implementing medical safety huddles — These short, virtual huddles are led by a huddle leader and occur on a weekly or once every two week basis. Each site will be adapting the Medical Safety Huddles for their context and workflow to specifically engage physicians.
  Arms: Medical Safety Huddles - Post-implementation

SUMMARY:
This quality improvement project will implement and evaluate the impact of physician-specific huddles, termed "medical safety huddles" on patient safety within four programs/sites at Sinai Health Systems, St. John's Rehab (Sunnybrook) and University Health Network.

ELIGIBILITY:
Inclusion criteria:

- Any staff physicians, residents or medical students working at the four programs/sites

Exclusion criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | 19 months
  We will examine whether the huddles impact the frequency and severity of adverse events experienced by patients. We will also determine if the huddles specifically impact certain types of adverse events in terms of frequency and severity. We will also perform analysis specific for each program/site.

SECONDARY OUTCOMES:
Process measure - Attendance rate | 15 months
  The number of physicians attending each huddle will be monitored to ensure the fidelity of implementation
Process measure - Safety issues | 15 months
  The type and number of safety issues brought up during huddles will be monitored on a monthly basis to ensure the fidelity of implementation
Process measure - Actions taken to address safety issues | 15 months
  The number of actions taken to address safety issues will be monitored on a monthly basis to ensure the fidelity of implementation

CONTACTS AND LOCATIONS:
Overall Officials: Meiqi Guo, MD, Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - St John's Rehab, Toronto, Ontario
  - Bridgepoint Active Health, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital - UHN, Toronto, Ontario1

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo M, Bayley M, Ye XY, Dunbar-Yaffe R, Fortin C, Go K, Macedo A, Matelski J, Mayo A, Pelc J, Robinson LR, Rotteau L, Wolfstadt J, Cram P, Linett L, Soong C. Impact of medical safety huddles on patient safety: a stepped-wedge cluster randomised study. BMJ Qual Saf. 2025 Sep 30:bmjqs-2025-019170. doi: 10.1136/bmjqs-2025-019170. Online ahead of print. PMID 41027730